CLINICAL TRIAL: NCT05878938
Title: Open-label Safety Study in Adults and Adolescents With Haemophilia A With and Without FVIII Inhibitors Switching Directly From Emicizumab Prophylaxis to NNC0365-3769 (Mim8) Prophylaxis
Brief Title: A Research Study Looking at How Safe it is to Switch From Emicizumab to Mim8 in People With Haemophilia A (FRONTIER 5)
Acronym: FRONTIER 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7769-4728; U1111-1281-9323 (Other: World Health Organization (WHO)); 2022-003053-66 (EudraCT Number)
Record Dates: First submitted 2023-05-12; First posted 2023-05-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia A; Haemophilia A With Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — protein phosphatase 4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NNC0365-3769 (Mim8) PPX (Experimental): Participants will receive Mim8 prophylaxis (PPX) subcutaneous (s.c.) injection using a prefilled fixed dose DV3407-C1 pen-injector.
  Interventions: Drug: NNC0365-3769 (Mim8) PPX

INTERVENTIONS:
Drug: NNC0365-3769 (Mim8) PPX — Participants will receive Mim8 PPX once-weekly dosing (QW), once every two weeks dosing (Q2W), or once-monthly dosing s.c. injection using a prefilled fixed dose DV3407-C1 pen-injector for 26 weeks.

SUMMARY:
This study is looking at how safe it is to switch from emicizumab to Mim8, in people with haemophilia A. Mim8 is a new medicine that is used to prevent bleeding episodes in people with haemophilia A. Mim8 works by replacing the function of the missing clotting factor VIII (FVIII). Mim8 will be injected under the skin using a pen-injector either once every week, once every two weeks or once every month. The participants will be trained in using the pen injector. The participants can choose themselves, in collaboration with the study doctor how often they get Mim8 in this study. When the participant will get their first Mim8 injection depends on their current treatment with emicizumab. The participants will get their first Mim8 injection at Visit 2. Participants will have between 6 and 27 Mim8 injections. The total number of injections participants will have depends on their dosing frequency. The study will last for about 6-12 months. While taking part in this study, there are some restrictions about what medicine participant can use. The study doctor will tell the participants more about this. In case the participants experience bleeds, these can be treated with additional haemostatic medicine as agreed with the study doctor. Female participants cannot take part if they are pregnant, breast-feeding or plan to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Male or female with diagnosis of congenital haemophilia A of any severity based on medical records.
3. Age 12 years or above at the time of signing the informed consent.
4. Participants treated with emicizumab once-weekly (QW), once every two weeks (Q2W), or once every four weeks (Q4W) according to the label for at least 8 weeks prior to screening.
5. Participants choosing to discontinue emicizumab treatment and switch to Mim8 QW, Q2W, or once-monthly (QM) treatment for 26 weeks from start of treatment (Visit 2).
6. Participant and/or caregiver willingness and ability to comply with scheduled visits and study procedures, including the completion of an electronic diary and patient-reported outcomes (PRO) questionnaires.

Exclusion Criteria:

1. Participation (i.e., signed informed consent) in any interventional, clinical study, with the exception of emicizumab, with receipt of the last dose within 8 weeks (or 5 half-lives of the investigational medicinal product [IMP], whichever is longer) before screening.
2. Any disorder, which in the investigator's opinion might jeopardise the participant's compliance with the protocol or safety, including ongoing Adverse Events (AEs) associated with emicizumab.
3. Previous participation in this study. Participation is defined as signed informed consent.
4. Known congenital or acquired coagulation disorders other than haemophilia A.
5. Previous or current thromboembolic disease or events (with the exception of previous catheter associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or risk of thromboembolic disease, as evaluated by investigator.
6. Neutralising antibodies towards emicizumab have been detected or, for patients adherent to emicizumab therapy, are suspected based on clinical and laboratory assessments.
7. Receipt of FVIII gene therapy at any time.
8. Ongoing or planned immune tolerance induction therapy.
9. Minor or major surgery planned to take place after screening and during the 26-week treatment period.
10. Known or suspected hypersensitivity to study intervention, related products, any constituents of the product or to other monoclonal antibodies.
11. Hepatic dysfunction defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) greater than (>) 3 times the upper limit combined with total bilirubin >1.5 times the upper limit measured at screening.
12. Renal impairment defined as estimated glomerular filtration rate (eGFR) lesser than or equal to (≤) 30 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) for serum creatinine measured at screening.
13. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive method.
14. Mental incapacity, unwillingness to cooperate, or a language barrier precluding adequate understanding and cooperation.
15. Other conditions (e.g. autoimmune disease) or laboratory abnormality that may increase risk of bleeding or thrombosis as evaluated by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | From Visit 2 (week 0) until week 26
  Measured as count of events.

SECONDARY OUTCOMES:
Device handling experience using the Hemophilia Device Handling and Preference Assessment (HDHPA) questionnaire | Visit 8 (after 26 weeks of treatment)
  Measured as percentage of participants. HDHPA measures device handling experience and device preference. The measure consists of 26 items that are reported individually. it is measures in units: Percentage of participants = the distribution of participant answers within each response category, for each of the 26 individual items.
Change in participants' treatment burden using the Hemophilia treatment experience measure (Hemo-TEM) total score | From Visit 2 (week 0) until end of treatment (up to 26 weeks)
  Measured as score points. Hemo-TEM measures treatment burden. The measure consists of 26 items yielding 5 domain scores and 1 total score. Domain scores (score range): Injection difficulties (0-100), physical impact (0-100), treatment bother (0-100), interference with daily life (0-100), and emotional impact (0-100). Total score ranges 0-100. Higher scores indicate greater treatment burden.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (36):
- United States (13):
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UC Denver Hemoph & Thrombo Ctr, Aurora, Colorado
  - St Joseph's Hospital Foundation, Tampa, Florida
  - Augusta Univ/Childrens Hosp-GA, Augusta, Georgia
  - Rush University Med. Cntr, Chicago, Illinois
  - University of Iowa_Iowa City, Iowa City, Iowa
  - Central Michigan University, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Univ Hosp Cleveland Med Ctr, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State MS Hershey Med Ctr, Hershey, Pennsylvania
  - Vanderbilt U Med Ctr_Nashville, Nashville, Tennessee
- Austria (2):
  - Universitätsklinik für Innere Medizin V, Innsbruck
  - AKH - Klin. Abt. f. Haematologie u. Haemostaseologie, Vienna
- Cliniques universitaires Saint-Luc - Service Hématologie, Brussels, Belgium
- McMaster University, Hamilton, Ontario, Canada
- Hospices Civils de Lyon- Hopital Louis Pradel-1, Bron, France
- Germany (2):
  - Vivantes Netzwerk für Gesundheit GmbH - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitätsklinikum Bonn - Institut für Experimentelle Hämatologie, Bonn
- Italy (4):
  - AOU Careggi Firenze, Florence, Tuscany
  - Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Rilievo Nazionale Santobono Pausilipon, Napoli
  - Azienda Ospedaliera Santobono Pausilipon - U.S.D. Centro Regionale Pediatrico Malattie della Coagulazione, Napoli
- Nara Medical University Hospital_Pediatrics, Nara, Japan
- Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng, South Africa
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- United Kingdom (6):
  - Belfast City Hospital, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Arthur Bloom Haemophilia Centre, Cardiff
  - Royal Free Haemophilia Comprehensive Care Center, London
  - Royal Free Haemophilia Comprehensive Care Centre, London
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com